CLINICAL TRIAL: NCT01103063
Title: A Phase 3, Open Label, Randomized, Comparative Study To Evaluate Azithromycin Plus Chloroquine And Sulfadoxine Plus Pyrimethamine Combinations For Intermittent Preventive Treatment Of Falciparum Malaria Infection In Pregnant Women In Africa
Brief Title: Evaluate Azithromycin Plus Chloroquine And Sulfadoxine Plus Pyrimethamine Combinations For Intermittent Preventive Treatment Of Falciparum Malaria Infection In Pregnant Women In Africa
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A0661158
Record Dates: First submitted 2010-04-07; First posted 2010-04-13 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-05

CONDITIONS: Intermittent Preventive Treatment In Pregnancy (IPTp)
Keywords: P. falciparum malaria; IPTp
MeSH Terms: interventions — Azithromycin; Chloroquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZCQ (Experimental): Azithromycin/chloroquine
  Interventions: Drug: Azithromycin plus chloroquine
- SP (Active Comparator): sulfadoxine-pyrimethamine (Fansidar)
  Interventions: Drug: sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Azithromycin plus chloroquine — combination tablet of 250mg azithromycin/155 chloroquine, Once daily PO for three days per treatment. There are total 3 treatments at 4-8 weeks intervals. The first treatment course will be administered during the second trimester (14-26 weeks of gestation as confirmed by ultrasound). The last treatment course should be given to subjects prior to or during 36 weeks of gestation.
  Arms: AZCQ
Drug: sulfadoxine-pyrimethamine — Fansidar tablet (500 mg sulfadoxine /25 mg pyrimethamine), once daily, PO, single dose per treatment. There are total 3 treatments at 4-8 weeks intervals. The first treatment course will be administered during the second trimester (14-26 weeks of gestation as confirmed by ultrasound). The last treatment course should be given to subjects prior to or during 36 weeks of gestation.
  Other Names: Fansidar
  Arms: SP

SUMMARY:
The primary objective is to establish superiority of AZCQ over SP in protective efficacy for IPTp as measured by the proportion of subjects with sub-optimal pregnancy outcome.

DETAILED DESCRIPTION:
After interim analysis of efficacy data by an External Data Monitoring Committee, this study was terminated. Investigators were notified on 22 Aug 2013. There were no safety concerns that led to this termination.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (all gravidae) with ≥14 and ≤26 weeks of gestational age (by ultrasound).
* Evidence of a personally signed and dated informed consent/assent document. Assent will be obtained from subjects <18 years of age.
* Subjects who are willing to and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Subjects who are available for follow up at delivery and on 28 days post delivery.

Exclusion Criteria:

* Age <16 years old or >35 years old.
* Multiple gestations as per the ultrasound at screening.
* Clinical symptoms of malaria.
* Hemoglobin < 8 g/dL (at enrollment).
* Any condition requiring hospitalization at enrollment.
* History of convulsions, hypertension, diabetes or any other chronic illness that may adversely affect fetal growth and viability.
* Inability to tolerate oral treatment in tablet form.
* Known allergy to the study drugs (azithromycin, chloroquine, and sulfadoxine-pyrimethamine) or to any macrolides or sulphonamides.
* Requirement to use medication during the study that might interfere with the evaluation of the study drug eg, trimethoprim-sulfamethoxazole use in subjects positive for HIV infection.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.
* Evidence of current obstetric complications that may adversely impact the pregnancy and/or fetal outcomes, including presence of congenital anomalies, placenta previa or abruption.
* Known severe Sickle Cell (SS) disease or Sickle Hemoglobin C (SC) anemia.
* Known family history of prolonged QT Syndrome, serious ventricular arrhythmia, or sudden cardiac death.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2891 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Benin (2):
  - Centre de Santé d'AHOUANSORI-AGUE, Cotonou, Benin
  - Hôpital Bethesda, Cotonou
- Siaya District Hospital, Siaya, Siaya County, Kenya
- Zomba Central Hospital, Zomba, Malawi
- Tanzania (4):
  - Teule Hospital, Muheza, Tanga
  - Nyamagana District Hospital, Mwanza, Tanzania
  - Bugando Medical Centre, Mwanza
  - Nyamagana District Hospital, c/o National Institute for Medical Research, Mwanza Centre, Mwanza
- Mulago Hospital Complex, Kampala, Uganda

REFERENCES:
- [Derived] Mtove G, Kimani J, Kisinza W, Makenga G, Mangesho P, Duparc S, Nakalembe M, Phiri KS, Orrico R, Rojo R, Vandenbroucke P. Multiple-level stakeholder engagement in malaria clinical trials: addressing the challenges of conducting clinical research in resource-limited settings. Trials. 2018 Mar 22;19(1):190. doi: 10.1186/s13063-018-2563-1. PMID 29566732
- [Derived] Kimani J, Phiri K, Kamiza S, Duparc S, Ayoub A, Rojo R, Robbins J, Orrico R, Vandenbroucke P. Efficacy and Safety of Azithromycin-Chloroquine versus Sulfadoxine-Pyrimethamine for Intermittent Preventive Treatment of Plasmodium falciparum Malaria Infection in Pregnant Women in Africa: An Open-Label, Randomized Trial. PLoS One. 2016 Jun 21;11(6):e0157045. doi: 10.1371/journal.pone.0157045. eCollection 2016. PMID 27326859
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661158&StudyName=Evaluate%20Azithromycin%20Plus%20Chloroquine%20And%20Sulfadoxine%20Plus%20Pyrimethamine%20Combinations%20For%20Intermittent%20Preventive%20Treatment%20Of%20Falciparum%20Malar

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open label, randomized, parallel group study screened a total of 3259 participants in 6 sites. A total of 2891 were treated either with azithromycin+chloroquine or sulfadoxine+pyrimethamine.
Pre-assignment Details: Pregnant women (all gravidae) with ≥14 and ≤26 weeks of gestational age were to be enrolled in this study. Approximately half of the participants were to be primigravidae and secundigravidae pregnant women since they had a higher risk for suboptimal pregnancy outcomes due to malaria.
Groups:
- Azithromycin + Chloroquine: The participants received 1000 mg Azithromycin (AZ) and 620 mg of Chloroquine (CQ) base (4 combination tablets of AZCQ with individual strength of 250 mg/155 mg), by mouth once daily for 3 days (Days 0, 1, 2) per treatment. There were a total of 3 treatments at 4-8 week intervals.
- Sulfadoxine + Pyrimethamine: The participants received sulfadoxine-pyrimethamine (SP) (Fansidar) treatment course: 1500 mg sulfadoxine and 75 mg pyrimethamine (3 fixed tablets of SP strength at 500 mg/25 mg), single oral dose on Day 0 of each treatment. There were a total of 3 treatments at 4-8 week intervals.
Period: Overall Study
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Started | 1446 | 1445
Completed | 969 | 1024
Not Completed | 477 | 421
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 68 | 51
Not completed — Withdrawal by Subject | 60 | 15
Not completed — Other | 16 | 11
Not completed — Protocol Violation | 1 | 0
Not completed — Study terminated by Sponsor | 326 | 342
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine | Total
Number analyzed (Participants) | 1446 | 1445 | 2891
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.3 (4.5) | 23.3 (4.6) | 23.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1446 | 1445 | 2891
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Participants With Sub-optimal Pregnancy Outcome in Intent-to-Treat (IIT) Population
Description: Adverse pregnancy outcomes were defined as live-borne neonate (singleton) with low birth weight (LBW) (<2,500 g), premature births (<37 weeks as confirmed by the Ballard score), abortion (≤28 weeks), still birth (>28 weeks), lost to follow-up prior to termination of pregnancy or delivery, or missing birth weight of the neonates.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants | 26.16 [23.89 to 28.43] | 23.67 [21.48 to 25.86]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; The 2-sided P-value tests the null hypothesis that the relative risk equals 1 (treatment group equality) versus not equal 1; Test type: Superiority or Other; p = 0.12237, Mantel Haenszel — Mantel-Haenszel estimate of the common relative risk is presented, adjusting for randomization strata. A relative risk less than 1 favors Azithromycin + Chloroquine treatment group (reduction in risk for the endpoint); Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.97 to 1.25], Standard Deviation 0.0647 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

2. Secondary Outcome: Percentage of Participants With Sub-optimal Pregnancy Outcome in Efficacy Analyzable Per Protocol (PP) Population
Description: Adverse pregnancy outcomes were defined as live-borne neonate (singleton) with LBW (<2,500g), premature births (<37 weeks as confirmed by the Ballard score), abortion (≤28 weeks), still birth (>28 weeks), lost to follow-up prior to termination of pregnancy or delivery, or missing birth weight of the neonates.
Time Frame: Approximately 40 weeks of gestational age
Population: Subset of ITT participants: outcome or withdrawal occurred on or before 8/27/2013 (date of study termination), compliant with study medication, birth weight measured on or before 7 days after birth if not already a failure, and did not switch to standard of care.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1089 | 1176
Percentage of Participants | 10.38 [8.57 to 12.19] | 10.12 [8.40 to 11.84]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.84117, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.80 to 1.31], Standard Deviation 0.1243 — The estimated risk ratio is presented along with its SE, with the SE on the log(e) scale

3. Secondary Outcome: Percentage of Neonates With LBW (<2500 g) in ITT Population
Description: LBW was defined as live birth weight <2500 g (up to and including 2499 g).
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Total live births.
Measure: Number (95% Confidence Interval); unit: Percentage of neonates
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1140 | 1190
Percentage of neonates | 5.01 [3.74 to 6.28] | 5.72 [4.40 to 7.04]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4428, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.62 to 1.23], Standard Deviation 0.1745 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

4. Secondary Outcome: Percentage of Neonates With LBW (<2500 g) in Efficacy Analyzable PP Population
Description: LBW was defined as live birth weight <2500 g (up to and including 2499 g).
Time Frame: Approximately 40 weeks of gestational age
Population: Subset of ITT participants: outcome or withdrawal occurred on or before 8/27/2013 (date of study termination), compliant with study medication, birth weight measured on or before 7 days after birth if not already a failure, and did not switch to standard of care. N=Total Live Births.
Measure: Number (95% Confidence Interval); unit: Percentage of neonates
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1041 | 1134
Percentage of neonates | 4.72 [3.43 to 6.01] | 5.21 [3.92 to 6.50]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6086, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.63 to 1.31], Standard Deviation 0.1882 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

5. Secondary Outcome: Percentage of Participants With Severe Maternal Anemia (Hemoglobin [Hb] <8 g/dL) at 36-38 Weeks of Gestation
Description: Severe maternal anemia was defined as Hb <8 g/dL.
Time Frame: At 36-38 weeks of gestation.
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of participants with Hb measurement at 36-38 weeks gestation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1222 | 1299
Percentage of participants | 1.80 [1.05 to 2.55] | 2.00 [1.24 to 2.76]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7035, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.51 to 1.57], Standard Deviation 0.2866 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

6. Secondary Outcome: Percentage of Participants With Maternal Anemia (Hb <11 g/dL) at 36-38 Weeks of Gestation
Description: Anemia was defined as Hb <11 g/dL.
Time Frame: At 36-38 weeks of gestation.
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1222 | 1299
Percentage of Participants | 50.57 [47.77 to 53.37] | 49.11 [46.39 to 51.83]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4605, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.95 to 1.11], Standard Deviation 0.0400 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

7. Secondary Outcome: Percentage of Participants With Placental Parasitemia at Delivery
Description: Participants with placental parasitemia at delivery were diagnosed using Placental blood smear at birth from participants who deliver at hospital.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of participants with placental parasite counts at delivery.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1019 | 1076
Percentage of participants | 5.30 [3.92 to 6.67] | 5.67 [4.29 to 7.05]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7105, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.65 to 1.33], Standard Deviation 0.1817 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

8. Secondary Outcome: Percentage of Participants With Placental Malaria at Delivery Based on Histology
Description: Participants positive for placental malaria at delivery were evaluated based on placental histology.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of participants with a histology parasite evaluation at delivery.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1040 | 1100
Percentage of participants | 4.81 [3.51 to 6.11] | 5.73 [4.36 to 7.10]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3468, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.59 to 1.21], Standard Deviation 0.1842 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

9. Secondary Outcome: Sexually Transmitted Infection (STI) Episodes Per Participant
Description: Number of episodes of sexually transmitted infection episodes per participant were noted. The STI's including Treponema pallidum, Neisseria gonorrhoeae, Chlamydia trachomatis, from first dose to delivery (diagnosis was based on clinical presentation and lab results).
Time Frame: Approximately 40 weeks of gestational age .
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of participants with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of episodes
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Number of episodes | 0.14 [0.11 to 0.16] | 0.19 [0.17 to 0.21]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; The 2-sided P-value tests the null hypothesis that the mean difference is 0 (treatment group equality) versus not equal 0; Test type: Superiority or Other; p = 0.0011, ANOVA — Analysis based on an ANOVA model with model terms for treatment group and randomization stratification variable. A negative mean difference between treatment groups favors Azithromycin + Chloroquine (reduction in number of STIs); Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.08 to -0.02], Standard Error of Mean 0.02

10. Secondary Outcome: Percentage of Participants With Sub-optimal Pregnancy Outcome Including Neonatal Death and Congenital Malformation
Description: Sub-optimal pregnancy outcome including neonatal deaths and congenital malformations, defined as any of the following: live-borne neonate (singleton) with low birth-weight (or LBW for short, defined as live birth weight <2,500g), premature birth (<37 weeks), abortion (≤28 weeks), still birth (>28 weeks), neonatal death, congenital malformation, lost to follow-up prior to termination of pregnancy or delivery, or missing birth weight of the neonates.
Time Frame: Approximately 40 weeks of gestational age.
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Total Outcomes.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants | 28.51 [26.18 to 30.84] | 26.51 [24.23 to 28.79]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2265, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.96 to 1.21], Standard Deviation 0.0604 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

11. Secondary Outcome: Change From Baseline to 36-38 Weeks of Gestation in Hb Concentration.
Description: Change from Baseline to 36-38 weeks of gestation in Hb concentration was noted.
Time Frame: Baseline, at 36-38 weeks of gestation.
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1221 | 1298
g/dL | 0.13 [0.05 to 0.21] | 0.27 [0.19 to 0.34]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0131, ANCOVA — Analysis based on an ANCOVA model with model terms for baseline value, treatment group and randomization stratification variable; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.24 to -0.03], Standard Error of Mean 0.05

12. Secondary Outcome: Percentage of Neonates With Congenital Abnormalities at Birth
Description: Neonates with congenital abnormalities at birth were noted.
Time Frame: Approximately 40 weeks of gestational age.
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of total live births.
Measure: Number (95% Confidence Interval); unit: Percentage of neonates
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1140 | 1190
Percentage of neonates | 2.19 [1.34 to 3.04] | 2.44 [1.56 to 3.31]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6978, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.53 to 1.53], Standard Deviation 0.2694 — The estimated risk ratio is presented along with its SE, with the SE on the log(e) scale

13. Secondary Outcome: Percentage of Perinatal or Neonatal Deaths
Description: Percentage of perinatal or neonatal deaths were noted.
Time Frame: Day 28 after delivery.
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percentage of neonates
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1140 | 1190
Percentage of neonates | 2.19 [1.34 to 3.04] | 1.85 [1.08 to 2.62]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6542, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.64 to 2.01], Standard Deviation 0.2908 — The estimated risk ratio is presented along with its SE, with the SE on the log(e) scale

14. Secondary Outcome: Birth Weight of Live Borne Neonate
Description: Birth weight of live borne neonates were calculated in grams.
Time Frame: Approximately 40 weeks of gestational age.
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 was considered the first dose of study medication), and who had a single fetus. N=Number of live births with available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1138 | 1188
grams | 3148.3 [3120 to 3176] | 3146.2 [3119 to 3174]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.9145, ANOVA — Analysis based on an ANOVA model with model terms for treatment group and randomization stratification variable; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-36.5 to 40.8], Standard Error of Mean 19.71

15. Secondary Outcome: Number of Episodes of Symptomatic Malaria Per Participant From First Intermittent Preventive Treatment of Falciparum Dose to Delivery
Description: This outcome measure determined if an episode of malaria started within the time period of first dose to delivery. Clinical episode of malaria was determined if the participant presented with clinical symptoms of malaria (fever >37.5°C, oral) and diagnosed (either by rapid diagnostic tests or microscopy) with malaria.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of episodes
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Number of episodes | 0.06 [0.04 to 0.08] | 0.13 [0.11 to 0.15]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Analysis based on an ANOVA model with model terms for treatment group and randomization stratification variable. A negative mean difference between treatment groups favors Azithromycin + Chloroquine (reduction in number of symptomatic malaria); Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.09 to -0.04], Standard Error of Mean 0.01

16. Secondary Outcome: Percentage of Participants Requiring Additional Treatment for Symptomatic Malaria From First Dose to Delivery
Description: This outcome measure evaluated the participants requiring additional treatments for malaria during the study period following the first dose (diagnosed based on clinical presentation and/or lab test results).
Time Frame: Approximately 40 weeks of gestational age
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants | 5.74 [4.54 to 6.94] | 10.52 [8.94 to 12.10]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.38 to 0.62], Standard Deviation 0.1221 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

17. Secondary Outcome: Percentage of Participants With Peripheral Parasitemia at 36-38 Weeks of Gestation
Description: This outcome measure evaluated the percentage of participants positive for peripheral parasitemia at 36-38 weeks of gestation. A participant was positive for parasitemia if the number of asexual parasites per μL was >0.
Time Frame: At 36-38 weeks of gestation
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N = Number of participants with peripheral blood smear parasite counts at 36-38 weeks of gestation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1069 | 1142
Percentage of participants | 2.71 [1.74 to 3.68] | 4.38 [3.19 to 5.57]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0360, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.39 to 0.97], Standard Deviation 0.2295 — The estimated risk ratio is presented along with its SE, with the SE on the log(e) scale

18. Secondary Outcome: Percentage of Participants With Peripheral Parasitemia at Delivery
Description: This outcome measure evaluated the percentage of participants positive for peripheral parasitemia at delivery. A participant was positive for parasitemia if the number of asexual parasites per μL was >0.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N = Number of participants with peripheral blood smear parasite counts at delivery.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1025 | 1086
Percentage of participants | 6.05 [4.59 to 7.51] | 7.46 [5.90 to 9.02]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1975, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.59 to 1.12], Standard Deviation 0.1630 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

19. Secondary Outcome: Percentage of Participants With Cord Blood Parasitemia at Delivery
Description: This outcome measure evaluated the percentage of participants positive for cord blood parasitemia at delivery. A participant was positive for parasitemia if the number of asexual parasites per μL was >0.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N = Number of participants with cord blood smear parasite counts at delivery.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1015 | 1072
Percentage of participants | 0.49 [0.06 to 0.92] | 0.75 [0.23 to 1.27]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4655, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.22 to 2.01], Standard Deviation 0.5675 — The estimated risk ratio is presented along with its SE, with the SE on the log(e) scale

20. Secondary Outcome: Percentage of Participants With Sexually Transmitted Infections From First Dose to 36-38 Weeks of Gestation
Description: Sexual transmitted disease included Treponema pallidum, Neisseria gonorrhoeae, and Chlamydia trachomatis infections. This was diagnosed based on clinical presentation prior to Week 36-38 and/or lab test results between Week 36-38.
Time Frame: Upto 36-38 weeks of gestation
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants | 12.32 [10.63 to 14.01] | 16.47 [14.56 to 18.38]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0016, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.62 to 0.90], Standard Deviation 0.0918 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

21. Secondary Outcome: Percentage of Participants With Chlamydia Trachomatis Infection at 36-38 Weeks of Gestation
Description: Participants positive for Chlamydia trachomatis infection was diagnosed based on laboratory result at 36-38 weeks of gestation. A vaginal swab was collected and PCR assay was used for analysis.
Time Frame: At 36-38 weeks of gestation
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N=Number of participants with lab test results at 36-38 weeks of gestation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 746 | 794
Percentage of participants | 1.47 [0.61 to 2.33] | 0.63 [0.08 to 1.18]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1113, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.34, 95% CI 2-sided [0.82 to 6.66], Standard Deviation 0.5338 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

22. Secondary Outcome: Percentage of Participants With Neisseria Gonorrhoeae Infection at 36-38 Weeks of Gestation
Description: Participants positive for Neisseria gonorrhoeae infection was diagnosed based on laboratory result at 36-38 weeks of gestation. A vaginal swab was collected and PCR assay was used for analysis.
Time Frame: At 36-38 weeks of gestation
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N=Number of participants with laboratory test results at 36-38 weeks of gestation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 746 | 794
Percentage of participants | 0.40 [0.00 to 0.85] | 1.64 [0.76 to 2.52]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0284, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.25, 95% CI 2-sided [0.07 to 0.86], Standard Deviation 0.6386 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

23. Secondary Outcome: Percentage of Participants With Treponema Pallidum Infection at 36-38 Weeks of Gestation
Description: Participants positive for Treponema pallidum infection was diagnosed based on laboratory result at 36-38 weeks of gestation. Treponema Pallidum particle Agglutination Assay was used.
Time Frame: At 36-38 weeks of gestation
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 751 | 797
Percentage of participants | 0.93 [0.24 to 1.62] | 2.01 [1.04 to 2.98]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0188, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.46, 95% CI 2-sided [0.24 to 0.88], Standard Deviation 0.3291 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

24. Secondary Outcome: Percentage of Participants With Trichomonas Vaginalis Infection at 36-38 Weeks of Gestation
Description: Participants positive for Trichomonas vaginalis infection was diagnosed based on laboratory result at 36-38 weeks of gestation. A vaginal swab was collected for the laboratory test.
Time Frame: At 36-38 weeks of gestation
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1068 | 1143
Percentage of participants | 8.24 [6.59 to 9.89] | 10.67 [8.88 to 12.46]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0527, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.59 to 1.00], Standard Deviation 0.1336 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

25. Secondary Outcome: Percentage of Participants With Bacterial Vaginosis Infection at 36-38 Weeks of Gestation.
Description: Bacterial vaginosis was diagnosed based on laboratory result at 36-38 weeks of gestation. A vaginal swab was collected for the Gram staining.
Time Frame: At 36-38 weeks of gestation
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 746 | 794
Percentage of participants | 8.58 [6.57 to 10.59] | 11.84 [9.59 to 14.09]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0384, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.54 to 0.98], Standard Deviation 0.1536 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

26. Secondary Outcome: Percentage of Neonates With Ophthalmia Neonatorum at Birth Period
Description: Ophthalmia neonatorum was diagnosed at birth. The laboratory diagnosis was performed among neonates with purulent discharge.
Time Frame: Approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N=Total live births.
Measure: Number (95% Confidence Interval); unit: Percentage of neonates
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1140 | 1190
Percentage of neonates | 0.35 [0.01 to 0.69] | 0.17 [0.00 to 0.40]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3942, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.09, 95% CI 2-sided [0.38 to 11.38], Standard Deviation 0.8648 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

27. Secondary Outcome: Percentage of Participants With Bacterial Infections Including Pneumonia and Other Lower Respiratory Tract Infections From First Dose to Delivery
Description: Participants positive for bacterial infections including other lower respiratory tract infections were measured anytime from first dose administration to delivery.
Time Frame: Up to approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N=Number of participants with available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants | 0.48 [0.13 to 0.84] | 1.25 [0.67 to 1.82]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0332, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.39, 95% CI 2-sided [0.16 to 0.93], Standard Deviation 0.4439 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

28. Secondary Outcome: Percentage of Participants With Pre-eclampsia From Week 20 to Delivery
Description: Pre-eclampsia was diagnosed as systolic blood pressure of at least 140 mmHg and/or diastolic blood pressure of at least 90 mmHg on two separate readings taken at least 4 hours apart and proteinuria at least 300 mg protein in a 24 hour urine collection.
Time Frame: From Week 20 to approximately 40 weeks of gestational age
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N= Number of participants with available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1440 | 1443
Percentage of participants | 0.63 [0.22 to 1.03] | 1.04 [0.51 to 1.55]
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2321, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.61, 95% CI 2-sided [0.27 to 1.38], Standard Deviation 0.4195 — The estimated risk ratio is presented along with its standard error (SE), with the SE on the log(e) scale

29. Secondary Outcome: Nasopharyngeal Swabs Positive for Macrolide Resistant Streptococcus Pneumoniae
Description: This outcome measure evaluated the Streptococcus pneumoniae sensitivity against macrolide antibiotics.
Time Frame: Visits 6 and 7
Population: ITT set was used which consisted of participants who were randomized, received at least one dose of study medication (Day 0 at Visit 1 is considered the first dose of study medication), and who had a single fetus. N=Number of participant with nasopharyngeal swabs isolating Streptococcus pneumoniae at the specified visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants
  Visit 6 (N = 8 and 17 respectively) | 0 | 11.76
  Visit 7 (N = 16 and 11 respectively) | 0 | 0
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; Statistical analysis for Visit 6 presented above; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = -11.76
Statistical Analysis 2: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; Statistical analysis for Visit 7 presented above; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = 0

30. Secondary Outcome: Nasopharyngeal Swabs Positive for Penicillin Resistant Streptococcus Pneumoniae
Description: This outcome measure evaluated the Streptococcus pneumoniae sensitivity against penicillin antibiotics.
Time Frame: Visits 6 and 7
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Azithromycin + Chloroquine | Sulfadoxine + Pyrimethamine
Number analyzed (Participants) | 1445 | 1445
Percentage of participants
  Visit 6 (N = 8 and 17 respectively) | 0 | 0
  Visit 7 (N = 16 and 11 respectively) | 0 | 0
Statistical Analysis 1: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; Statistical analysis for Visit 6 presented above; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = 0
Statistical Analysis 2: Comparison: Azithromycin + Chloroquine vs Sulfadoxine + Pyrimethamine; Statistical analysis for Visit 7 presented above; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Mean Difference (Final Values) = 0

ADVERSE EVENTS:
Time Frame: Up to Visit 7 (6 months post last dose). Includes data up to 35 days after last dose of study drug for mothers (treatment emergent), and includes all data for neonates.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. Some events are seen only in neonates (e.g neonatal malformation/anomalies, LBW etc.) and are not expected in mothers and vice versa. Such events are designated as 'zero' in the respective 'familial status- neonate/mother' in the below table.
Groups:
- Mother (Azithromycin + Chloroquine): The participants received 1000 mg Azithromycin (AZ) and 620 mg of Chloroquine (CQ) base (4 combination tablets of AZCQ with individual strength of 250 mg/155 mg), by mouth once daily for 3 days (Days 0, 1, 2) per treatment. There were a total of 3 treatments at 4-8 week intervals.
- Mother (Sulfadoxine + Pyrimethamine): The participants received sulfadoxine-pyrimethamine (SP) (Fansidar) treatment course: 1500 mg sulfadoxine and 75 mg pyrimethamine (3 fixed tablets of SP strength at 500 mg/25 mg), single oral dose on Day 0 of each treatment. There were a total of 3 treatments at 4-8 week intervals.
- Neonate (Azithromycin + Chloroquine): Live births of participants who received 1000 mg Azithromycin (AZ) and 620 mg of Chloroquine (CQ) base (4 combination tablets of AZCQ with individual strength of 250 mg/155 mg), by mouth once daily for 3 days (Days 0, 1, 2) per treatment. There were a total of 3 treatments at 4-8 week intervals.
- Neonate (Sulfadoxine + Pyrimethamine): Live births of participants who received sulfadoxine-pyrimethamine (SP) (Fansidar) treatment course: 1500 mg sulfadoxine and 75 mg pyrimethamine (3 fixed tablets of SP strength at 500 mg/25 mg), single oral dose on Day 0 of each treatment. There were a total of 3 treatments at 4-8 week intervals.
Arm/Group | Mother (Azithromycin + Chloroquine) | Mother (Sulfadoxine + Pyrimethamine) | Neonate (Azithromycin + Chloroquine) | Neonate (Sulfadoxine + Pyrimethamine)
Serious Adverse Events (participants affected / at risk) | 65/1446 | 42/1445 | 101/1149 | 104/1196
Other Adverse Events (participants affected / at risk) | 1177/1446 | 888/1445 | 301/1149 | 326/1196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mother (Azithromycin + Chloroquine) (N=1446) | Mother (Sulfadoxine + Pyrimethamine) (N=1445) | Neonate (Azithromycin + Chloroquine) (N=1149) | Neonate (Sulfadoxine + Pyrimethamine) (N=1196)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 2
Haemorrhagic disease of newborn (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0
Anal atresia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Cerebellar hypoplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital hand malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Congenital malaria (Congenital, familial and genetic disorders) | 0 | 0 | 3 | 2
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 2
Cystic lymphangioma (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Exomphalos (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 2 | 1
Microgenia (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 16 | 21
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectourethral fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Death neonatal (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 2 | 9 | 2 | 3
Meningitis (Infections and infestations) | 1 | 0 | 1 | 1
Neonatal infection (Infections and infestations) | 0 | 0 | 5 | 4
Pneumonia (Infections and infestations) | 1 | 1 | 9 | 10
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 3
Sepsis neonatal (Infections and infestations) | 0 | 0 | 11 | 13
Skin bacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Apgar score low (Investigations) | 0 | 0 | 1 | 1
HIV test positive (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 0 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 4 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 7 | 1 | 0 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 9 | 10
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Placental infarction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 | 5 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 17 | 12
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 7 | 5 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 4 | 4 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 4 | 3 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 5 | 7 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 | 3 | 0 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal vessel disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 9
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 5
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mother (Azithromycin + Chloroquine) (N=1446) | Mother (Sulfadoxine + Pyrimethamine) (N=1445) | Neonate (Azithromycin + Chloroquine) (N=1149) | Neonate (Sulfadoxine + Pyrimethamine) (N=1196)
Anaemia (Blood and lymphatic system disorders) | 205 | 192 | 21 | 14
Vision blurred (Eye disorders) | 145 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 123 | 50 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 120 | 36 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 50 | 45 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 205 | 14 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 15 | 0 | 0
Gastritis (Gastrointestinal disorders) | 23 | 7 | 0 | 0
Nausea (Gastrointestinal disorders) | 216 | 58 | 0 | 0
Vomiting (Gastrointestinal disorders) | 650 | 96 | 0 | 0
Asthenia (General disorders) | 239 | 40 | 0 | 0
Fatigue (General disorders) | 81 | 22 | 0 | 0
Pyrexia (General disorders) | 10 | 26 | 40 | 28
Conjunctivitis (Infections and infestations) | 0 | 0 | 15 | 10
Gastroenteritis (Infections and infestations) | 44 | 21 | 48 | 37
Infection parasitic (Infections and infestations) | 14 | 18 | 0 | 0
Malaria (Infections and infestations) | 49 | 121 | 37 | 37
Pneumonia (Infections and infestations) | 0 | 0 | 34 | 25
Sepsis (Infections and infestations) | 0 | 0 | 18 | 9
Sepsis neonatal (Infections and infestations) | 0 | 0 | 21 | 21
Trichomoniasis (Infections and infestations) | 58 | 55 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 127 | 153 | 125 | 116
Urinary tract infection (Infections and infestations) | 105 | 115 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 75 | 60 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 19 | 20 | 0 | 0
White blood cells urine positive (Investigations) | 149 | 162 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 44 | 11 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 29 | 0 | 0
Dizziness (Nervous system disorders) | 460 | 84 | 0 | 0
Headache (Nervous system disorders) | 300 | 219 | 0 | 0
Somnolence (Nervous system disorders) | 38 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 29 | 39
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 28 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 10 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 46 | 23 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 22 | 8 | 0 | 0

LIMITATIONS AND CAVEATS:
This program was terminated by Pfizer based on the results of the pre-planned interim analysis for this pivotal study. The interim analysis showed no benefit of the study drug (AZCQ) compared to standard of care (SP).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.